CLINICAL TRIAL: NCT00992849
Title: Topical/Subconjunctival Injection of Bevacizumab(Avastin) for the Treatment of Corneal Neovascularization
Brief Title: Bevacizumab for the Treatment of Corneal Neovascularization
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Ching-Hsi Hsiao, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-0918C
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Corneal Neovascularization
Keywords: Corneal neovascularization; bevacizumab
MeSH Terms: conditions — Corneal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Arm type to experimental based on single group assignment. Bevacizumab (trade name Avastin, Genentech/Roche) is a humanized monoclonal antibody that recognises and blocks vascular endothelial growth factor (VEGF).VEGF is a chemical signal that stimulates the growth of new blood vessels.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Topical 10 mg/cc or subconjunctival 2.5 mg/0.1cc
  Other Names: Avastin

SUMMARY:
The purpose of the current study is to assess the efficacy and safety of the inhibitory effect of bevacizumab (Avastin) with different routes including topical and subconjunctival application on corneal neovascularization in the human eyes.

DETAILED DESCRIPTION:
The compassionate off-label use of bevacizumab as well as the potential risks, benefits, and adverse effects of this medication are discussed extensively with each patient. To further minimize systemic absorption, silicone punctual plugs are placed in the lower eyelids. One group of patients apply topical bevacizumab, 1.0%(10mg/ml), 4 times of day. The other group of patients received subconjunctival injection of bevacizumab(2.5mg/0.1ml) once. The patients are examined at 1day, 1week, 2weeks, 3weeks, and 1month, then monthly till the corneal neovascularization are gone or reduced to some degrees. Best-corrected visual acuity, slip-lamp examination, tonometry, external photography, pachymetry, specular microscopy (if possible), and systemic blood pressure are completed at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Significant unilateral or bilateral corneal neovascularization that extending over the limbus at least 2mm.
* The underlying etiologies that caused corneal neovascularization included post penetrating keratoplasty (PKP), ocular surface reconstruction , trauma, infectious or non-infectious corneal ulcer.
* Corneal neovascularization induced lipid keratopathy, corneal edema, or irregular corneal surface. The best-corrected visual acuity was less than 20/25.
* Post-PSP or ocular surface reconstruction corneal neovascularization that had no associated lipid keratopathy, no corneal edema, or corneal irregularity. But the neovascularization was highly possible to cause graft rejection.
* The corneal neovascularization was refractory to other medical treatment.
* The patient had received PKP or other corneal surgeries mort than half a year ago and was not in the acute post-operation phase.
* The patient had no active endophthalmitis, glaucoma with uncontrolled intraocular pressure, or vitreoretinal diseases.
* The patient signed inform consent to have regular follow up and treatment.

Exclusion Criteria:

* The neovascularization had clinical improvement three months before the first injection.
* The lipid keratopathy had clinical improvement three months before the first injection.
* The patient that suspected to have poor visual outcome or had already been light sense negative Glaucoma patient that had uncontrolled intraocular pressure.
* Poor corneal epithelialization.
* Patient that had systemic disease which was not suitable for bevacizumab use.
* Pregnant patient.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Regression of corneal neovascularization | 6 months

SECONDARY OUTCOMES:
visual acuity, lipid keratopathy, side effect | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsi Hsiao, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan